CLINICAL TRIAL: NCT06803355
Title: The Value of Systemic Inflammation Markers in Differentiating Congenital Pneumonia From TTN in Neonates
Brief Title: Comparison of Congenital Pneumonia and Transient Tachypnea of the Newborn
Status: Completed | Type: Observational
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Ceren Akdag, Assistant Doctor, Dr. Behcet Uz Children's Hospital
Other Study IDs: BU-PEDS-CA-01
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Congenital Pneumonia; Transient Tachypnea of the Newborn
Keywords: Biomarker; Newborn; Inflammation
MeSH Terms: conditions — Transient Tachypnea of the Newborn; Inflammation | interventions — Blood Cell Count; Blood Culture; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Biospecimen Retention: Samples Without DNA — Complete blood count, blood smear test, C- reactive protein, blood culture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- congenital pneumonia: patients diagnosed with congenital pneumonia
  Interventions: Diagnostic Test: complete blood count, CRP, blood smear test, blood culture, chest X- ray
- transient tachypnea of the newborn: patients diagnosed with transient tachypnea of the newborn
  Interventions: Diagnostic Test: complete blood count, CRP, blood smear test, blood culture, chest X- ray

INTERVENTIONS:
Diagnostic Test: complete blood count, CRP, blood smear test, blood culture, chest X- ray — Inflammation markers obtained from all cases will be evaluated and used to differentiate between transient tachypnea of the newborn and congenital pneumonia.

SUMMARY:
Accurate and timely differentiation between transient tachypnea of the newborn (TTN) and congenital pneumonia is essential in neonatal care, as it facilitates prompt initiation of appropriate treatment, reduces the risk of complications, and minimizes inappropriate antibiotic use. This study aims to assess the clinical utility of inflammatory markers, including the Systemic Immune-Inflammation Index (SII) and the Systemic Immune-Response Index (SIRI), in distinguishing TTN from congenital pneumonia in neonates. In scenarios where conventional diagnostic methods prove insufficient, these indices may offer clinicians a reliable and objective diagnostic approach, thereby optimizing antibiotic stewardship and reducing the duration of hospitalization.

DETAILED DESCRIPTION:
Patients admitted to the Neonatal Intensive Care Unit of Dr. Behçet Uz Children's Hospital for respiratory distress will be analyzed.

The following data will be recorded in the "case report form" for each patient: age, gender,Score for Neonatal Acute Physiology- Perinatal Extension-II (SNAPPE-II), birth weight (SGA/LGA), mode of delivery (elective/emergency C-section and vaginal delivery), gravidity, parity, maternal age, maternal comorbidities (GDM, preeclampsia/eclampsia, hypothyroidism, chorioamnionitis, urinary tract infection, asthma, obesity, epilepsy), presence of premature rupture of membranes or fever, sibling history, low APGAR score (<7), leukocyte count, neutrophil count, lymphocyte count, platelet count, monocyte count, aspartate transferase (AST), C-reactive protein (CRP), blood smear test, blood culture, tracheal aspirate culture, antibiotics used and their duration, chest X-ray findings, length of hospital stay, onset and duration of oxygen therapy and method of administration, need for mechanical ventilation, and morbidity and mortality status.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born at ≥37 weeks of gestation,
* Admitted within the first 24 hours after birth with respiratory distress

Exclusion Criteria:

* Congenital anomalies
* Genetic syndromes
* Diagnosis of sepsis
* Patients without informed consent

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population includes term neonates (≥37 weeks of gestation) diagnosed with either transient tachypnea of the newborn (TTN) or congenital pneumonia. All patients are evaluated within the first 24 hours postnatally (0-24 hours). Only neonates admitted to the neonatal intensive care unit (NICU) for respiratory distress are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Differentiation of TTN and congenital pneumonia using systemic immune-inflammation index (SII) | within the first 24 hours postnatally
  The Systemic Immune-Inflammation Index (SII) is a biomarker derived from neutrophil count, lymphocyte count, and platelet count. It has been shown to increase proportionally with the degree of inflammation.
Differentiation of TTN and congenital pneumonia using systemic inflammatory response index (SIRI) | within the first 24 hours postnatally
  The Systemic Inflammatory Response Index (SIRI) is a biomarker derived from neutrophil count, lymphocyte count, and monocyte count. It has been shown to increase proportionally with the degree of inflammation.

SECONDARY OUTCOMES:
Effectiveness of Inflammatory Markers in Differentiating TTN and Congenital Pneumonia | within the first 24 hours postnatally
  inflammatory markers such as neutrophil-lymphocyte ratio (NLR), pan-immune-inflammation value (PIV) , platelet-lymphocyte ratio (PLR), AST to platelet ratio index (APRI) typically increase during inflammation, while lymphocyte- monocyte ratio (LMR) generally decreases.
Differentiation of TTN and congenital pneumonia using C Reaktive Protein | 24 hours postnatally
  CRP has been shown to increase proportionally with the degree of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Şebnem Çalkavur, MD, Study Director — Dr. Behcet Uz Children's Hospital
Locations (1):
- Dr. Behçet Uz Children's Hospital, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao L, Liu X, Sun T, Zhang Y, Bao T, Cheng H, Tian Z. Predictive and Diagnostic Values of Systemic Inflammatory Indices in Bronchopulmonary Dysplasia. Children (Basel). 2023 Dec 25;11(1):24. doi: 10.3390/children11010024. PMID 38255338
- [Background] Kumar A, Bhat BV. Epidemiology of respiratory distress of newborns. Indian J Pediatr. 1996 Jan-Feb;63(1):93-8. doi: 10.1007/BF02823875. PMID 10829971